CLINICAL TRIAL: NCT01172054
Title: A Phase I Escalating Dose Ranging Study to Evaluate the Safety and Immunogenicity of the VAX128 A, B, and C Novel H1N1 Influenza Vaccine Constructs in Healthy Adults 18-49 Years of Age and in Community Living Adults ≥65 Years of Age
Brief Title: Comparative Safety and Immunogenicity of VAX128A, VAC128B and VAX128C Novel H1N1 Influenza Vaccine in Healthy Adults
Acronym: VAX128-01
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VaxInnate Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: VAX128-01
Record Dates: First submitted 2010-07-26; First posted 2010-07-29 (Estimated); Last update posted 2012-07-31 (Estimated); Status verified 2012-07

CONDITIONS: Influenza
Keywords: influenza vaccine recombinant
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- VAX128 (Experimental): Novel H1N1 Influenza vaccine
  Interventions: Biological: VAX128
- Placebo (Placebo Comparator): one IM injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VAX128 — one IM injection
  Other Names: STF2.HA1 CA07
  Arms: VAX128
Biological: Placebo — One IM injection
  Arms: Placebo

SUMMARY:
This is a multicenter, escalating dose-ranging study to assess the safety, reactogenicity and immunogenicity of 3 different novel H1N1 influenza vaccine constructs delivered i.m. as a single dose vaccination on day 0.

DETAILED DESCRIPTION:
VAX128-01 is a first in human study of three inactivated recombinant novel H1N1 influenza vaccines, designated VAX128 A, B and C. The purpose of the study is to compare the safety and immunogenicity of the three vaccines through a range of doses and to select one of the vaccines for further testing in phase II studies. We plan to assess the safety and immunogenicity in a dose escalating study. The study will enroll up to 100 healthy young adults (18-49 years) and 100 healthy adults than age 65 years. We are including the older adults in this phase 1 study because we have found that the elderly tolerated a vaccine similar to one of the candidates, VAX128A, better than young adults, but required a higher vaccine dose to achieve a similar antibody response. Nevertheless, because we are testing two other constructs (VAX128B and C), we will be making the conservative assumptions that the safety and immunogenicity data coming from the young adults will not predict the results in the elderly. Therefore, we will begin the study in the young adults and after the first three dose levels have been tested we will begin testing in the older adults. In this study we plan to enroll up to 100 young adults and up to 100 adults 65 years and older. The young adults will be most likely enrolled at one clinical site and the older adults will be enrolled at another clinical site. We plan to enroll a cohort of 10 young adults and 10 older adults every week. Each cohort will consist of 3 subjects to receive one of the three vaccines (9 subjects total) and one subject in each cohort will receive placebo. Dosing for the next cohort will be based on a two day assessment period after vaccination. The main part of the study will be conducted over 28 days and there will be two follow up phone calls at 6 months and one year.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female aged 18 - 49 years or >= 65 years
* Give written informed consent
* Females have a negative urine test for pregnancy before vaccination and use birth control during 28 day study period
* Willing to receive the unlicensed (VAX128) vaccine given as an i.m. injection
* Willing to provide multiple blood specimens collected by venipuncture

Exclusion Criteria:

* Chronic illness that would interfere with the subject's participation in the study or interpretation of the study results.
* Impaired immune responsiveness
* Received drugs effecting the immunity
* Received or plan to receive a nonstudy vaccine within 30 days prior to vaccination and during the study, including licensed influenza vaccines.
* History of anaphylactic type reaction to injected vaccines.
* History of drug abuse in the year prior to screening.
* History of Guillain-Barré Syndrome.
* Receipt or donation of blood products
* Acute disease within 72 hours prior to vaccination
* History of heart or lung disease
* Has other conditions that might interfere with study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Safety | 28 days
  Assess safety, reactogenicity and tolerability. Symptoms will be collected from the memory aid and from the information collected at the clinic visits. All symptoms will be graded according to severity. Response to vaccine will be categorized as local (arm pain, redness, bruising etc) or systemic (headache, muscle aches, fatigue, etc) symptoms. Laboratory tests such as CRP, WBC, LFTs and cytokines collected before and after vaccination will also be analyzed. We will compare the types and severity of symptoms and laboratory results based on vaccine construct or placebo.

SECONDARY OUTCOMES:
Immunogenicity | 28 days
  To assess serm immune response, sera collected at Day 0 (pre-vaccination), 7, 14 and 28 will be analyzed for HAI, serum IgG anti-HA by ELISA and serum IgG anti-flagellin by ELISA. The geometric mean, seroconversion and seroprotection rates will be determined.

CONTACTS AND LOCATIONS:
Overall Officials: David N Taylor, MD, Study Director — VaxInnate Corporation
Locations (2):
- United States (2):
  - Miami Research Associates, Miami, Florida
  - Johnson County Clin-Trials, Lenexa, Kansas

REFERENCES:
- [Derived] Taylor DN, Treanor JJ, Sheldon EA, Johnson C, Umlauf S, Song L, Kavita U, Liu G, Tussey L, Ozer K, Hofstaetter T, Shaw A. Development of VAX128, a recombinant hemagglutinin (HA) influenza-flagellin fusion vaccine with improved safety and immune response. Vaccine. 2012 Aug 24;30(39):5761-9. doi: 10.1016/j.vaccine.2012.06.086. Epub 2012 Jul 11. PMID 22796139